CLINICAL TRIAL: NCT04681716
Title: Effect of Mobilization With and Without ELDOA in Lumber Radiculopathy
Brief Title: Effects of ELDOA in Lumber Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aqua Medical Services (Pvt) Ltd (Industry)
Responsible Party: Principal Investigator, Mir Arif Hussain, Assistant professor, Aqua Medical Services (Pvt) Ltd
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00129 M.jibran
Record Dates: First submitted 2020-11-27; First posted 2020-12-23 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Lumbar Radiculopathy
Keywords: ELDOA; mobilization; lumber radiculopathy; NPRS; ODI
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ELDOA GROUP (Active Comparator): ELDOA position was instructed to this group
  Interventions: Other: ELDOA
- CONVENTIONAL PHYSIOTHERAPY (Experimental): Hot pack,TENS and mobalization was given in this group
  Interventions: Other: CONVENTIONAL PHYSIOTHERAPY

INTERVENTIONS:
Other: ELDOA — For Spinal Segment L4-L5 and L5-S1 proper ELDOA position was instructed to the experiment group patients.ELDOA stands for Elongation Longitudinaux Avec Decoaption Osteo Articulaire, or LOADS (Longitudinal Osteo-articular De-coaptation Stretching). ... They can be described as fascial stretch that localizes tension at the level of a specific spinal segmental.
  Arms: ELDOA GROUP
Other: CONVENTIONAL PHYSIOTHERAPY — Transcutaneous Electrical Nerve Stimulation (TENS):
  120Z dual channel TENS unit made in Japan was used in the research. Electrodes of TENS were placed on lumbar region and TENS was given for 15 minutes on Constant mode. Intensity was adjusted according to patient's comfort.
  Hot pack was applied on the lumbar region for 10 - 15 minutes.Lumbar Mobilization (CPA) was given on spinous process of L1- L5 vertebrae and L5-S1. For every session given 3 sets of 10 repetitions of each lumbar vertebra was performed.
  Arms: CONVENTIONAL PHYSIOTHERAPY

SUMMARY:
ELDOA is the most beneficial intervention treating for lumbar pathologies such as radiculopathy. This study was a randomized control trial in which data was collected from Riphah Rehabilitation and Research Centre and Pakistan Railway Hospital-IIMCT. Purposive sampling technique was used for data collection. Research data was recorded by using prescribed validated questionnaire, NPRS and ODI. After taking consent from patients, patients were divided randomly in two groups through lottery method. Group A was treated with ELDOA and mobilization, group B was treated with only mobilization. It was observed that both groups showed improvement but ELDOA group showed more significant results.

DETAILED DESCRIPTION:
ELDOA is the most beneficial intervention treating for lumbar pathologies such as radiculopathy. ELDOA is defined as (Etirements Longitudinaux avec Decoaptation Osteo-Articulaire), it's a collective series of programmed group of exercises which are created to show remarkable improvements and to focus on healthy posture and a renowned French osteopath Guy Voyer, D.O also emphasized on development of spinal health. ELDOA are specially designed programmed exercises it regain the place of membranous fascia, soft structures such as muscles , cord like structures such as ligaments and tendons of a gliding surfaces like joints and vertebral body in their primary positions to the specified joints or spinal segmental areas.Musicians should be importantly acknowledge that: the shear forces arises due to repetition of movements because of activities of daily living , practicing and performances which lies down soft structure such as tissues, resulting in default posture and faulty alignment which after prolong time headed towards painful symptoms and dysfunction of normal structures. As in between the joints ELDOA forms adequate space in joints and a marked improvement is observed with in mechanics of gliding services such as joints, flow of blood also increases , with this pressure on intervertebral segmental discs also decreases ,inter-segmental hydration is regained, hyper tonicity in muscles occur, alertness, adrenal gland hormonal and equilibrium of metabolism occurs, also the tensions created by the myofascial like structures get to normal state, decrease in pain perception, progression toward ideal posture, different stages of sleep is markedly improved, and the sensation of being healthy is also gained. How does it occur? In physiotherapy common practice ELDOA assumed postures produces proper spacing in joints physically, it also allows aqua fluid to re-enter , moreover it provides early healing and cushioning to the structures, it also prepares the neuronal circuits to get adopt by nervous system and readjust the newly assumed positioning of the gliding joints. With time it also improves and also eliminates painful symptoms along with physical abnormalities.The advantages of regular clinical ELDOA practices are proved to be very effective and has significant effect on improving living standards , one perception of living, and how ones feels , it also show improvement in joint functioning and mobility and increases the performance through working on its source. Despite of one's mobility and strength, flexibility, the protocols affecting the progression factors and least almost zero impact of EDOLA exercises makes it possible to be followed by everyone and are fully effective for health. ELDOA is being used 2.8% worldwide. Its prevalence is increasing rapidly because of its positive immediate effects.ELDOA is a combination of static exercises of strengthening and stretching that includes myofascial compartment and it helps to decompress the affected joints along with it also functionalizes the facial compartment. From the advantages it includes limitation beyond shaping the intrinsic muscles of spinal column and providing more strength and stability along with it decreases the risk of accidental injury functionalizing spinal segmental disc from effect of decompression forces, it also shape's the stretched muscles that are suspensory soft structures such as muscles and organ tissues that are connective in nature. Moreover EDOLA showed not only marked improvement but also enhanced adaptive postural health and also maintain posture of IS health. The spinal canal is arranged as house of exiting nerves that nourish our organs and the structures such as connective tissues that deeply suspends into the organs and increases their functioning and they are intact with the spinal column.ELDOA has significant effect on fluids and tissues it creates normalization, cellular level decompression and traction. When abnormal dysfunction occur proprioception, nerves, membranous structures such as fascia, ligaments and soft structures like muscle, organs are normalize by implantation of EDOLA and through this undergoing functioning of various systems such as of endocrine, hormonal changes and even activities of nervous system can also be notified. ELDOA also has significant effect globally body various systems and also locally allocating them back into harmony range and it also utilizes micro movements which further uproot macro functioning. In common practice it is observed that implementation of EDLOA has significant effect on normal digestion and absorption action, reproductive and geriatric function, improved sleep, decrease palpitations in heart along with decreases issues related to backache , moreover for an ordinary client having health related back issues it is not unusual for him to undergo the process of ELDOA.

The main criteria of this descriptive study is to analyze the effectiveness of interventional treatments such as ELDOA and graded mobilization techniques in comparison, Both interventions are utilize to treat radiculopathy issues of lumbar segment which arises because of disc issues such as herniation, emphasis is on the development of beneficial treatment and efficient enough to proceed toward no surgical procedures method for affected persons in physiotherapy sciences to treat them with problems of radiculopathy of lumbar segmental area may arise due to disc health issues like herniation and to create such effective method which ensures more better instantly and long lasting results of ELDOA in treating the patients with radiculopathy of lumbar segmental area which arises due to disc herniation. a baseball player say that ELDOA's on the other hand allow for natural spinal and joint decompression which also allows for larger range of motion (the more open the spine the more a hitter is able to rotate and create hip separation which allows for increased power production), freedom of movement, and ultimately more athleticism.The object is to create a position that targets a specific intervertebral level, by creating a decoarctation between a fixed point means the inferior vertebra, and a mobile point the superior vertebra , which the object maintains through his/her own myofascial tension of a particular articular chain and result in the targeted intervertebral decoarctation. The technique of ELDOA define as step wise is as:1)Create a position that targets a specific intervertebral level,2)Creating a decoarctation between a fixed point (the inferior vertebra) and a mobile point (the superior vertebra).3)Maintains through his or her own myofascial tension of a particular articular chain and results in the targeted intervertebral decoarctation.4)The clinician monitors the position to provide objective feedback and coaches and encourages the patient.5)The clinician uses verbal, visual, and touch cues and works to use these cues Simultaneously. 6)Stack tensions and engage the whole body 7)Work in a holistic or multilevel way .8)Not to hold the breath or to strain with breathing but as far as possible to encourage a relaxed, "natural" diaphragmatic breathing.9)Once the patient is in the position, the clinician needs to palpate at the target articular level and cue the patient with "fine tuning" until he/she feels the decoaptation movement at the target level. 10)Patients to travel around inside their body and learn to fine tune themselves.11)The therapist has to work on progressions before the final position can be obtained by the patient.In daily routine PT cannot practice ELDOA to treat their patients that's why very few researches are seen on ELDOA in Pakistan. Evidence shows that ELDOA has significant results on musculoskeletal disorders; it can help in treating patients. This study will explains that ELDOA is very much effective in treating lumbar radiculopathy and it can improve their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Radicular pain radiates into the lower extremity

  * Positive response of at least 4 of the following test
  * SLR test
  * Limited ROM
  * Valsalva maneuver
  * Lumbar Compression Test
  * Deep tendon reflexes (knee and ankle jerk).

Exclusion Criteria:

* Inflammatory Arthritis, Mass occupied lesion, Fracture, piriformis syndrome.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-08-27 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | immediately after intervention
  The Numeric Pain Rating Scale (NPRS) is a one-dimensional measure of pain intensity in individuals. in which patient selects a number (0-10) from a horizontal line that best reflects the intensity of their pain, with 0 representing no pain and 10 representing pain as bad as one can imagine or worst pain imaginable. The number that the patient point to on the scale to rate their pain intensity is recorded. Higher scores indicate greater pain intensity. NPRS was used and patients were asked to rate their pain before the first treatment session and then at the end of last treatment session.

SECONDARY OUTCOMES:
Oswestry Disability Index (Modified ODI) for Low Back Pain | immediately after intervention
  The Oswestry Disability Index (Modified ODI) is a self-rating outcome tool for low back pain disability and it is also recognized as the Oswestry Disability Questionnaire for Low Back Pain. In the year 1980, Fairbank et al, introduced ODI, it provides information about low back pain disability and its effects on the potential to handle daily life activities. The test is considered as the 'gold standard' of low back functional outcome. ODI consists of 10 sections indicating functional status in daily activities i.e. regarding pain, personal care, weight lifting, walking, sitting, standing, sleeping, social life, traveling and employment /homemaking. Every section has 6 options scored from 0 to 5 with 0 being normal and 5 being the worst outcome possible. Patient is instructed to mark one best possible answer. The total score for questionnaire is 50. After calculating the individual score percentage is taken by dividing it with total score i.e. 50 and multiplying by 100

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Ghafoor Sajjad,, PHD*, Principal Investigator — Shifa Tameer e milat University
Locations (1):
- Aqua research Center, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kelsey JL. An epidemiological study of the relationship between occupations and acute herniated lumbar intervertebral discs. Int J Epidemiol. 1975 Sep;4(3):197-205. doi: 10.1093/ije/4.3.197. PMID 1184269
- [Background] O'Sullivan MG, Connolly AE, Buckley TF. Recurrent lumbar disc protrusion. Br J Neurosurg. 1990;4(4):319-25. doi: 10.3109/02688699008992741. PMID 2222878
- [Background] Pynsent FJ. Oswestry Low Back Pain Disability Questionnaire 1980 [cited 2016 2 August]; Available from: http://www.rehab.msu.edu/_files/_docs/Oswestry_Low_Back_Disability.pdf.
- [Background] Haegg O. Oswestry Disability Index. Encyclopedia of Pain: Springer; 2013. p. 2559-62.
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Hammer WI. Functional soft-tissue examination and treatment by manual methods: Jones & Bartlett Learning; 2007.
- [Background] Morre N, Planat C. Sur trois granites des sondages de Marchenoir, Boissy-sur-Saint-Yon et Courgent de la partie occidentale du bassin de Paris. Bulletin de la Sociéte geologique de France. 1964;5(3):358-62.
- [Background] McCarroll JR, Miller JM, Ritter MA. Lumbar spondylolysis and spondylolisthesis in college football players. A prospective study. Am J Sports Med. 1986 Sep-Oct;14(5):404-6. doi: 10.1177/036354658601400513. PMID 3777317
- [Background] Lee RY, Evans JH. Loads in the lumbar spine during traction therapy. Aust J Physiother. 2001;47(2):102-8. doi: 10.1016/s0004-9514(14)60301-9. PMID 11552865